CLINICAL TRIAL: NCT00496132
Title: An Open-Label, Multicenter, Phase I/II Trial of the Safety of Escalating Doses of PRO131921 in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia Who Have Been Treated With a Purine Nucleoside Analogue-Containing Regimen
Brief Title: A Trial of the Safety of Escalating Doses of PRO131921 in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACO4198g
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; Leukemia; Lymph
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — PRO131921 monoclonal antibody

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PRO131921

INTERVENTIONS:
Drug: PRO131921 — Escalating doses by IV infusion

SUMMARY:
This is an open-label, multicenter, Phase I/II study of the safety of escalating doses of single-agent PRO131921 in patients with chronic lymphocytic leukemia (CLL) who have relapsed after or were refractory to treatment with a purine nucleoside analogue-containing regimen. The trial will enroll in two phases: a Phase I dose-escalation portion and a Phase II expanded treatment cohort, with enrollment of additional patients in order to expand safety experience and collect preliminary anti-leukemia activity data.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of histologically confirmed B-cell CLL
* Relapsed or refractory CLL with history of prior treatment with purine nucleoside analogue-containing regimen
* Eligible for treatment of their CLL based on criteria adapted from the National Cancer Institute-Working Group (NCI-WG) Response Criteria for CLL
* For patients of reproductive potential (males and females), use of a reliable means of contraception
* For females of childbearing potential, a negative serum pregnancy test

Exclusion Criteria:

* Prior use of anti-CD20 monoclonal antibody therapy (other than rituximab)
* Prior use of any non-CD20 targeted monoclonal antibody therapy within 6 months of enrollment
* Current or recent CLL treatment
* History of severe allergic or anaphylactic reactions to human, humanized, chimeric, or murine monoclonal antibodies
* Evidence of acute/active autoimmune hemolytic anemia or other autoimmune complications of CLL
* Use of hematopoietic growth factors or RBC and/or platelet transfusions
* Evidence of significant uncontrolled concomitant diseases, such as cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine, or gastrointestinal disorders
* Evidence of myelodysplasia or myelodysplastic changes on bone marrow examination
* History of cancer other than CLL)
* Known active bacterial, viral, fungal, mycobacterial, or other infection or any major episode of infection requiring hospitalization or treatment with IV antibiotics or oral antibiotics
* A major episode of infection requiring hospitalization or treatment with IV antimicrobials within 4 weeks of screening or oral antimicrobials within 2 weeks of screening
* Positive hepatitis B or C serology
* Positive human immunodeficiency virus (HIV) serology
* Active cytomegalovirus (CMV) disease by antigen or polymerase chain reaction testing
* Pregnancy or lactation
* CNS leukemia
* Recent major surgery, other than diagnostic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-08-27 (Actual); Primary Completion 2009-06-17 (Actual); Study Completion 2009-06-17 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities and adverse events | Length of study

SECONDARY OUTCOMES:
Pharmacokinetic parameters; CD19-positive B-cell counts | Length of study
Overall response rate and progression-free survival (Phase II only) | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Bill Ho, M.D., Study Director — Genentech, Inc.